CLINICAL TRIAL: NCT05455333
Title: Clinical Interest of a Genetic Diagnosis in Early Infant Epilepsy, Paraclinical and Therapeutic Management, and Psychological Impact of Families
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8609
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Early Infant Epilepsy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Sends and returns questionnaires to families.

SUMMARY:
To determine the paraclinical and therapeutic interest of genetic diagnosis in early onset epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Children aged ≤ 12 years,
* hospitalized or followed at the Hautepierre Hospital of the University Hospitals of Strasbourg for primary epilepsy having started in the first 5 months of life, from 2010 to 2021.

Exclusion Criteria:

- Children with secondary epilepsy (with infection trauma)

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged ≤ 12 years, hospitalized or followed at the Hautepierre Hospital of the University Hospitals of Strasbourg for primary epilepsy having started in the first 5 months of life, from 2010 to 2021.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of event densities | 4 month
  The frequency of events (crises, going to the emergency room, hospitalizations) before and after genetic diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Génétique Médicale IGMA - Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided